CLINICAL TRIAL: NCT02624219
Title: A Phase I Randomized, Double-Blind, Controlled Trial in Healthy Adults to Assess the Safety, Reactogenicity, and Immunogenicity of a Monovalent Inactivated Influenza A/H5N8 Virus Vaccine Administered Intramuscularly at Different Dosages Given With or Without AS03 or MF59 Adjuvants
Brief Title: H5N8 Mix and Match With or Without AS03 or MF59 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15-0064; HHSN272201300020I
Record Dates: First submitted 2015-11-25; First posted 2015-12-08 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Avian Influenza; Influenza
Keywords: A/H5N8; AS03; Controlled; Double-Blind; Immunogenicity; Inactivated; Influenza; MF59; Monovalent; Randomized; Reactogenicity; Safety; Trial; Vaccine
MeSH Terms: conditions — Influenza in Birds; Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Group 1 (Experimental): N = 55 receive 7.5 mcg A/H5N8 + AS03 on Day 1, 22
  Interventions: Drug: AS03; Biological: Monovalent Influenza A/H5N8 vaccine
- Group 2 (Experimental): N = 55 receive 7.5 mcg A/H5N8 + MF59 on Day 1, 22
  Interventions: Drug: MF59 adjuvant; Biological: Monovalent Influenza A/H5N8 vaccine
- Group 3 (Experimental): N = 55 receive 15 mcg A/H5N8 unadjuvanted on Day 1, 22
  Interventions: Biological: Monovalent Influenza A/H5N8 vaccine
- Group 4 (Experimental): N = 55 receive 15 mcg A/H5N8 + AS03 on Day 1, 22
  Interventions: Drug: AS03; Biological: Monovalent Influenza A/H5N8 vaccine
- Group 5 (Experimental): N = 55 receive 15 mcg A/H5N8 + MF59 on Day 1, 22
  Interventions: Drug: MF59 adjuvant; Biological: Monovalent Influenza A/H5N8 vaccine

INTERVENTIONS:
Drug: AS03 — AS03 oil-in-water emulsion adjuvant.
  Arms: Group 1; Group 4
Drug: MF59 adjuvant — Microfluoridized adjuvant 59 (MF59) is an oil-in-water emulsion.
  Arms: Group 2; Group 5
Biological: Monovalent Influenza A/H5N8 vaccine — Monovalent inactivated influenza A/H5N8 virus vaccine for IM injection. prepared from influenza virus propagated in chicken egg fluid using seed virus prepared from the candidate vaccine virus (CVV), influenza virus A/gyrfalcon/Washington/41088-6/2014(H5N8)-PR8-IDCDC-RG43A (abbreviated as IDCDC-RG43A).

SUMMARY:
This is a Phase I randomized, double-blind, controlled trial in 275 males and non-pregnant females, 19 to 64 years old, inclusive, who are in good health and meet all eligibility criteria. This clinical trial is designed to assess the safety, reactogenicity, and immunogenicity of a monovalent inactivated influenza A/H5N8 virus vaccine manufactured by bioCSL administered at different dosages (7.5 or 15 mcg of HA/0.5 mL dose) given with or without AS03 or MF59 adjuvants manufactured by GlaxoSmithKline Biologicals and Novartis Vaccines and Diagnostics, respectively.

DETAILED DESCRIPTION:
This is a Phase I randomized, double-blind, controlled trial in 275 males and non-pregnant females, 19 to 64 years old, inclusive, who are in good health and meet all eligibility criteria which include screening hematology, chemistry and erythrocyte sedimentation rate (ESR) laboratory evaluations. This clinical trial is designed to assess the safety, reactogenicity, and immunogenicity of a monovalent inactivated influenza A/H5N8 virus vaccine manufactured by bioCSL administered at different dosages (7.5 or 15 mcg of HA/0.5 mL dose) given with or without AS03 or MF59 adjuvants manufactured by GlaxoSmithKline Biologicals and Novartis Vaccines and Diagnostics, respectively. The primary objectives of this study is to assess 1) the safety and reactogenicity of a monovalent inactivated influenza A/H5N8 virus vaccine and 2) the serum hemagglutination inhibition (HAI) and neutralizing (Neut) antibody responses to a monovalent inactivated influenza A/H5N8 virus vaccine following receipt of two doses administered intramuscularly at different dosages (7.5 or 15 mcg of HA/0.5 mL dose) given with or without AS03 or MF59 approximately 21 days apart. The secondary objectives of this study are to 1) assess study vaccine-related unsolicited non-serious adverse events following receipt of two doses of a monovalent inactivated influenza A/H5N8 virus vaccine, 2) assess medically attended adverse events (MAAEs) including new-onset chronic medical conditions and immune-mediated or auto-inflammatory adverse events of special interest following receipt of two doses of a monovalent inactivated influenza A/H5N8 virus vaccine, and 3) assess the serum HAI and Neut antibody responses to a monovalent inactivated influenza A/H5N8 virus vaccine following receipt of one dose administered intramuscularly at different dosages (7.5 or 15 mcg of HA/0.5 mL dose) given with or without AS03 or MF59. This study will span approximately 24 months. Subject participation duration will span approximately 13 months.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to initiation of any study procedures. 2. Are able to understand and comply with planned study procedures and be available for all study visits. 3. Are males or non-pregnant females, 19 to 64 years old, inclusive. 4. Are in good health. Note: As determined by medical history and physical examination to evaluate acute or currently ongoing chronic medical diagnoses or conditions, defined as those that have been present for at least 90 days, that would affect the assessment of the safety of subjects or the immunogenicity of study vaccinations. Chronic medical diagnoses or conditions should be stable for the last 60 days. This includes no change in chronic prescription medication, dose, or frequency as a result of deterioration of the chronic medical diagnosis or condition in the 60 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site principal investigator or appropriate sub-investigator, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening of medical diagnosis or condition. Similarly, medication changes subsequent to enrollment and study vaccination are acceptable provided there was no deterioration in the subject's chronic medical condition that necessitated a medication change, and there is no additional risk to the subject or interference with the evaluation of responses to study vaccination. Note: Topical, nasal, and inhaled medications (with the exception of inhaled corticosteroids as outlined in the Subject Exclusion Criteria (see Section 5.1.2)), herbals, vitamins, and supplements are permitted. 5. Oral temperature is less than 100.0°F. 6. Pulse is 50 to 115 bpm, inclusive. 7. Systolic blood pressure is 85 to 150 mmHg, inclusive. 8. Diastolic blood pressure is 55 to 95 mmHg, inclusive. 9. Erythrocyte sedimentation rate (ESR) is less than 30 mm per hour. 10. Alanine aminotransferase (ALT) is less than 44 IU/L for females or is less than 61 IU/L for males. 11. Creatinine is less than 1.11 mg/dL for females or is less than 1.38 mg/dL for males. 12. White blood cells (WBC) are greater than 3.9 x10^3/µL and less than 10.6 x10^3/µL. 13. Hemoglobin (Hgb) is greater than 11.4 g/dL for females or is greater than 12.4 g/dL for males. 14. Platelets are greater than 139 x10^3/µL and less than 416 x10^3/µL. 15. Total bilirubin is less than 1.3 mg/dL. 16. Women of childbearing potential* must use an acceptable contraception method** from 30 days before the first study vaccination until 60 days after the last study vaccination. *Not sterilized via tubal ligation, bilateral oophorectomy, hysterectomy or successful Essure® placement with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or <1 year of the last menses if menopausal. **Includes, but is not limited to, non-male sexual relationships, abstinence from sexual intercourse with a male partner, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more prior to the subject receiving the first study vaccination, barrier methods such as condoms or diaphragms with spermicide or foam, effective intrauterine devices, NuvaRing®, and licensed hormonal methods such as implants, injectables or oral contraceptives ("the pill"). 17. Women of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to study vaccination.

Exclusion Criteria:

1. Have an acute illness*, as determined by the site principal investigator or appropriate sub-investigator, within 72 hours prior to study vaccination. *An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site principal investigator or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol. 2. Have any medical disease or condition that, in the opinion of the site principal investigator or appropriate sub-investigator, is a contraindication to study participation**. **Including acute or chronic medical disease or condition, defined as persisting for at least 90 days, that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial. 3. Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to study vaccination. 4. Have known active neoplastic disease or a history of any hematologic malignancy. Non-melanoma skin cancers are permitted. 5. Have known human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection. 6. Have known hypersensitivity or allergy to eggs, egg or chicken protein, squalene-based adjuvants, or other components of the study vaccine. 7. Have a history of severe reactions following previous immunization with licensed or unlicensed influenza virus vaccines. 8. Have a personal or family history of narcolepsy. 9. Have a history of Guillain-Barré syndrome. 10. Have a history of convulsions or encephalomyelitis within 90 days prior to study vaccination. 11. Have a history of autoimmune or auto-inflammatory disease***. ***Including, but not limited to, autoimmune or auto-inflammaory processes resulting in neuralgia, paresthesia, neuritis, neuroinflammatory diseases, vasculitis, clotting disorders, dermatitis, arthritis, thyroiditis, hypothyroidism, hyperthyroidism, or muscle, liver, or kidney disease. Refer as well to the list of AESIs. 12. Have a history of alcohol or drug abuse within 5 years prior to study vaccination. 13. Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations. 14. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 10 years prior to study vaccination. 15. Have taken oral or parenteral (including intraarticular) corticosteroids of any dose within 30 days prior to study vaccination. 16. Have taken high-dose inhaled corticosteroids within 30 days prior to study vaccination. High-dose defined as >840 mcg/day of beclomethasone dipropionate CFC or equivalent. 17. Received a licensed live vaccine within 30 days prior to the first study vaccination, or plan to receive a licensed live vaccine within 30 days before or after each study vaccination. 18. Received a licensed inactivated vaccine within 14 days prior to the first study vaccination, or plan to receive a licensed inactivated vaccine within 14 days before or after each study vaccination. 19. Received immunoglobulin or other blood products (with exception of Rho D immunoglobulin) within 90 days prior to study vaccination. 20. Received an experimental agent7 within 30 days prior to the first study vaccination, or expect to receive an experimental agent8 during the 13-month trial-reporting period. 7Including vaccine, drug, biologic, device, blood product, or medication. 8Other than from participation in this trial. 21. Are participating or plan to participate in another clinical trial with an interventional agent**** that will be received during the 13-month trial-reporting period. ****Including licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication. 22. Prior participation in a clinical trial of influenza A/H5 vaccine***** or have a history of influenza A/H5 virus actual or potential exposure or infection prior to the first study vaccination. *****And assigned to a group receiving influenza A/H5 vaccine, does not apply to documented placebo recipients. 23. Occupational exposure to or substantial direct physical contact (Note) with birds in the past year or during the 21 days after each study vaccination. Note: Casual contact with birds at petting zoos, county or state fairs, or having pet birds does not exclude subjects from study participation. 24. Female subjects who are breastfeeding or plan to breastfeed at any given time from the first study vaccination until 30 days after the last study vaccination. 25. Plan to travel outside the US (continental US, Hawaii, and Alaska) within 21 days after each study vaccination.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 276 (Actual)
Dates: Start 2016-08-16 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Titers of serum HAI and Neut antibodies against the A/H5N8 antigen contained in the study vaccine | Approximately 21 days after the second study vaccination
Occurrence of clinical safety laboratory adverse events | Day 22-30
Occurrence of clinical safety laboratory adverse events | Day 1-9
Occurrence of solicited injection site and systemic reactogenicity events | Day 1-9
Occurrence of solicited injection site and systemic reactogenicity events | Day 22-30
Occurrence of study vaccine-related serious adverse events | Day 1-387
Percentage of subjects achieving a serum HAI antibody titer of 1:40 or greater against the A/H5N8 antigen contained in the study vaccine | Approximately 21 days after the second study vaccination
Percentage of subjects achieving a serum Neut antibody titer of 1:40 or greater against the A/H5N8 antigen contained in the study vaccine | Approximately 21 days after the second study vaccination
Percentage of subjects achieving HAI seroconversion against the A/H5N8 antigen contained in the study vaccine | Approximately 21 days after the second study vaccination
Percentage of subjects achieving Neut seroconversion against the A/H5N8 antigen contained in the study vaccine | Approximately 21 days after the second study vaccination

SECONDARY OUTCOMES:
Geometric Mean Titers of serum HAI and Neut antibodies against the A/H5N8 antigen contained in the study vaccine | At baseline and approximately 8, 21 and 29 days after the first study vaccination
Occurrence of MAAEs including new-onset chronic medical conditions and immune-mediated or auto-inflammatory AESIs | Day 1-387
Occurrence of study vaccine-related unsolicited non-serious adverse events after vaccination 1 | Day 1-22
Occurrence of study vaccine-related unsolicited non-serious adverse events after vaccination 2 | Day 22-43
Percentage of subjects achieving HAI seroconversion against the A/H5N8 antigen contained in the study vaccine | At approximately 8, 21 and 29 days after the first study vaccination
Percentage of subjects achieving Neut seroconversion against the A/H5N8 antigen contained in the study vaccine | At approximately 8, 21 and 29 days after the first study vaccination
Percentage of subjects achieving serum HAI and Neut antibody titers of 1:40 or greater against the A/H5N8 antigen contained in the study vaccine | At baseline and approximately 8, 21 and 29 days after the first study vaccination

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Iowa - Vaccine Research and Education Unit, Iowa City, Iowa
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas